CLINICAL TRIAL: NCT02367846
Title: The Effect of Oral vs. Non-oral Contraceptive Therapy on Bone Turnover Using 41Ca Methodology
Brief Title: Assessing the Impact of Contraceptives on Bone Health Using 41Ca
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Mary Jane DeSouza, Professor of Kinesiology and Physiology, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000464
Record Dates: First submitted 2015-01-27; First posted 2015-02-20 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Other Disorders of Bone Development and Growth
Keywords: Calcium Tracer; Oral Contraceptives; Contraceptive Vaginal Ring; Impact of contraceptives on bone health using 41Ca
MeSH Terms: interventions — Contraceptives, Oral, Combined; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined Oral Contraceptive (COC) (Experimental): We are testing the effects of a COC (Apri (Reclipsen); 30 µg EE, 150 µg desogestrel). On the first day of the intervention, the participants randomized to COC will begin taking the pill. One pill will be ingested orally at the same time each day for days 1-49 of the intervention. Pills ingested during days 1-21 and during days 29-49 will be active tablets. Pills ingested on days 22-28 will be tablets without active ingredients. Each participant in the COC group will ingest a pill from the first pack each day for the first 28 days then begin the second pack. If a participant is unable to collect a 24-h urine sample on day 49, she will take active tablets from the third pill pack until she has collected the 24-h urine sample.
  Interventions: Drug: Combined Oral Contraceptive (COC)
- Contraceptive Vaginal Ring (CVR) (Experimental): We are testing the effects of the vaginal ring (Nuva Ring; 15 µg/d EE, 120 µg/d etonogestrel). When randomized to CVR, participants will insert the contraceptive ring into their vagina . The ring will be worn during weeks 1-3, and again during weeks 5-7. During week 4, no ring will be worn to allow for withdrawal bleeding. If a participant is unable to collect a 24-h urine sample on day 49, they will insert a third ring which will remain in the vagina until she has collected a 24-h urine sample.
  Interventions: Drug: Contraceptive Vaginal Ring (CVR)

INTERVENTIONS:
Drug: Combined Oral Contraceptive (COC) — The proposed study is a preclinical, multi-site trial comparing the short-term effects of oral vs. non-oral ethinyl estradiol on net bone calcium balance. A prospective crossover study with repeated measures and a simple random assignment will be used to test the effects of 49 days of COC use on bone metabolism using 41Ca to determine net bone calcium balance. Subjects will be randomized to receive COC during either the first or second intervention period.
  Other Names: Apri (Reclipsen)
  Arms: Combined Oral Contraceptive (COC)
Drug: Contraceptive Vaginal Ring (CVR) — The proposed study is a preclinical, multi-site trial comparing the short-term effects of oral vs. non-oral ethinyl estradiol on net bone calcium balance. A prospective crossover study with repeated measures and a simple random assignment will be used to test the effects of 49 days of CVR use on bone metabolism using 41Ca to determine net bone calcium balance. Subjects will be randomized to receive CVR during either the first or second intervention period.
  Other Names: Nuva Ring
  Arms: Contraceptive Vaginal Ring (CVR)

SUMMARY:
This preclinical randomized crossover study will examine the effects of oral versus non-oral contraceptive therapy on bone turnover in young exercising women. In an effort to expose the route-dependent effects of oral versus non-oral contraceptive therapy on bone turnover, the investigators will examine 1) the effects of ethinyl estradiol on bone calcium balance using the 41Ca technology and 2) the underlying physiological mechanisms associated with the effects of oral versus non-oral contraceptive therapy on net bone calcium balance.

DETAILED DESCRIPTION:
This study is a preclinical, multi-site study (Penn State University and Purdue University) that will determine whether the negative effects of combined oral contraceptive (COC) therapy on bone turnover are dependent on the route of administration such that an attenuation of these effects is observed when a comparable dose of non-oral contraceptive therapy, such as vaginal contraceptive (CVR) therapy is also tested. Millions of women use COC therapy for birth control purposes or regulation of menstrual cycles. CVR therapy is a relatively new FDA-approved contraceptive alternative to COC. The purpose of the proposed project is to investigate whether oral ethinyl estradiol (EE) may negatively impair bone turnover when compared to vaginally-administered EE in young physically-active women.

A novel calcium tracer technology suitable to rapidly assess changes in net bone calcium balance in a small sample size will be applied to evaluate the effects of COC and CVR therapy on bone turnover. The radioisotope Calcium-41 (41Ca) demonstrates increased sensitivity when compared to dual x-ray absorptiometry (DXA) and increased specificity for bone mineralization and precision when compared to biochemical markers of bone turnover. This study will be the first study to examine how the route of estrogen administration affects bone turnover in young physically active women by assessing changes in net bone calcium balance with different forms of contraceptive therapy.

The overall purpose of this study is to explore the effects of oral versus vaginal contraceptive therapy on bone turnover in young exercising women using 41Ca technology. In an effort to expose the route-dependent effects of oral versus non-oral contraceptive therapy on bone turnover, the investigators will examine 1) the effects of ethinyl estradiol on bone calcium balance using the 41Ca technology and 2) the underlying physiological mechanisms associated with the effects of oral versus vaginal contraceptive therapy on net bone calcium balance.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18-25 yrs
3. BMI 18-29 kg/m2
4. Non-smoking
5. Willing to refrain from using hormonal contraceptives for the equilibration + baseline period of the study (~150 days)
6. Availability to frequently visit the laboratory in the next 12 months
7. Not currently pregnant nor intending to become pregnant in the next 12 months
8. Not lactating
9. No apparent metabolic, endocrine, musculoskeletal, or severe psychiatric disease
10. Willing to maintain consistent exercise (aerobic, weight-bearing) and dietary habits during pre-intervention and intervention periods
11. Willing to refrain from supplements other than those provided by study staff in the next 12 months
12. Variable physical activity acceptable, but mode must be primarily weight bearing
13. At least 9 menses in the past 12 months

Exclusion Criteria:

1. Non-weight bearing exercise as primary mode of physical activity
2. Resistance exercise training (≥ 2 times 30 minutes per week of resistance exercise)
3. Complete seasonal change of impact mode of physical activity
4. Known or suspected metabolic or endocrine disease
5. Smoking
6. Pregnant
7. Currently consuming large amounts of soy products
8. Current clinical eating disorder or other axis 1 psychiatric disorder or bipolar disorders
9. Oral or hormonal contraceptive use in the last 6 months
10. Hyperparathyroidism
11. Liver or renal disease
12. Evidence of malabsorption or skeletal disorder
13. Thyroid abnormalities (controlled hypothyroidism acceptable)
14. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDS)
15. Taking medications known to have interactions with oral or vaginal contraceptive therapy
16. Other Exclusion Criteria proposed by the World Health Organization COC Contraindications (Grossman et al., 2011).

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in 41Ca:Ca ratio | 49 days of contraceptive therapy
  Changes in the 41Ca:Ca ratio in 24-h urine samples measured every 10-14 days during and after oral and non-oral contraceptive therapy as determined by Accelerometer Mass Spectrometry

SECONDARY OUTCOMES:
Changes in serum concentrations of insulin-like growth factor-1 (IGF-1), IGF-binding proteins (IGFBP-1, IGFBP-3), and acid labile subunit (ALS) | 49 days of contraceptive therapy
  Changes in fasting serum concentrations of IGF-1, IGFBP-1, IGFBP-3, and ALS after oral and non-oral contraceptive therapy
Changes in serum concentrations of markers of bone formation and bone resorption | 49 days of contraceptive therapy
  Changes in fasting serum concentrations of markers of bone formation (osteocalcin, P1NP) and bone resorption (CTx) after oral and non-oral contraceptive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane De Souza, PhD, Principal Investigator — Penn State University
Locations (1):
- Women's Health and Exercise Laboratories, The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Grossman D, White K, Hopkins K, Amastae J, Shedlin M, Potter JE. Contraindications to combined oral contraceptives among over-the-counter compared with prescription users. Obstet Gynecol. 2011 Mar;117(3):558-565. doi: 10.1097/AOG.0b013e31820b0244. PMID 21343758
- [Background] Lee WH, Wastney ME, Jackson GS, Martin BR, Weaver CM. Interpretation of 41Ca data using compartmental modeling in post-menopausal women. Anal Bioanal Chem. 2011 Feb;399(4):1613-22. doi: 10.1007/s00216-010-4454-5. Epub 2010 Dec 9. PMID 21152905
- [Background] Weaver CM, Martin BR, Jackson GS, McCabe GP, Nolan JR, McCabe LD, Barnes S, Reinwald S, Boris ME, Peacock M. Antiresorptive effects of phytoestrogen supplements compared with estradiol or risedronate in postmenopausal women using (41)Ca methodology. J Clin Endocrinol Metab. 2009 Oct;94(10):3798-805. doi: 10.1210/jc.2009-0332. Epub 2009 Jul 7. PMID 19584189
- [Background] Denk E, Hillegonds D, Vogel J, Synal A, Geppert C, Wendt K, Fattinger K, Hennessy C, Berglund M, Hurrell RF, Walczyk T. Labeling the human skeleton with 41Ca to assess changes in bone calcium metabolism. Anal Bioanal Chem. 2006 Nov;386(6):1587-602. doi: 10.1007/s00216-006-0795-5. Epub 2006 Oct 11. PMID 17033771